CLINICAL TRIAL: NCT04188158
Title: Analysis of the Effectiveness of Neoadjuvant Chemotherapy in the Treatment of Colon Cancer Locally Advanced
Brief Title: Analysis of the Effectiveness of Neoadjuvant Chemotherapy in the Treatment of Colon Cancer Locally Advanced (ELECLA)
Acronym: ELECLA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, Dr. Jorge Arredondo, PRINCIPAL INVESTIGATOR, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nº AEMPS: 16-0553; 2016-002970-10 (EudraCT Number)
Record Dates: First submitted 2019-11-25; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Locally Advanced Colon Cancer
MeSH Terms: interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: * Intervention Group: Neoadjuvant chemotherapy + surgery + adjuvant chemotherapy
  * Control group: surgery + adjuvant chemotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 3 cycles XELOX + Surgery+ 5 cycles XELOX
  Interventions: Combination Product: CAPECITABINE AND OXALIPLATIN
- Control group (Other): Surgery + 8 cycles XELOX
  Interventions: Combination Product: CAPECITABINE AND OXALIPLATIN

INTERVENTIONS:
Combination Product: CAPECITABINE AND OXALIPLATIN — Intervention Group: Neoadjuvant chemotherapy ( 3 cycles Capecitabine and oxaliplatin) + surgery + adjuvant chemotherapy (5 cycles Capecitabine and oxaliplatin)

SUMMARY:
Effectiveness analysis of neoadjuvant chemotherapy in the treatment of locally advanced colon cancer. ELECLA trial

DETAILED DESCRIPTION:
Participants in this study selected patients according to homogeneous inclusion criteria and will be treated either with a uniform protocol of neoadjuvant chemotherapy, surgery and complementary chemotherapy (intervention group), or with the standard scheme of postoperative surgery and chemotherapy (control group ). All patients will be studied basally through clinical examinations and radiological and endoscopic tests usually used to reach the diagnosis of Locally Advanced Colon Cancer . In the group of patients receiving neoadjuvant treatment, the CT scan will be repeated after the completion of preoperative chemotherapy to restage the disease and quantify the degree of tumor response.

Finally, the project tries to determine whether the neoadjuvant treatment scheme increases disease-free survival (SLE) at 2 and 5 years and overall survival (OS) at 5 years. Likewise, the toxicity derived from chemotherapy treatment and perioperative morbidity and mortality will be analyzed to evaluate the feasibility and safety of the therapeutic procedure. The rate of completion of chemotherapy in both groups will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* CLINICS

  1. Histological confirmation of colon adenocarcinoma.
  2. Patients of both sexes with age over 18 years.
  3. Good general condition of the patient (Karnofsky> 60% or ECOG (Eastern Cooperative Oncology Group) <2).
  4. Analytical at the time of inclusion with figures of Hemoglobin> 10 g / dL; Leukocytes> 3.0 109 / L, Platelets> 100,000, Glomerular Filtration> 50 ml / min and Total Bilirubin <25 micromol / l.
  5. Absence of contraindication for chemotherapy.
  6. Acceptance and signature of the Informed Consent.
* OF IMAGE

  1. Radiological signs, evaluated by CT, of T4 or T3 tumor infiltration> 5 mm of transmural invasion.
  2. With or without lymph node involvement by CT.
  3. No metastatic involvement in other organs (M0).
  4. Radiologically resectable disease. REFERENCES TO THE TREATMENT

  <!-- -->

  1. That they will undergo elective surgery with curative intent (R0).

Exclusion Criteria:

* 1. Important comorbidity, uncontrolled angina or a history of acute myocardial infarction in the last 6 months.

  2. Personal history of another malignancy in the last 5 years, with the exception of melanoma.

  3. Uncontrolled infection 4. Pregnancy or lactation. 5. Peripheral neuropathy> grade 1. 6. Rectum cancer (<15 cm of the anal margin or below peritoneal reflection). 7. Presence of distant metastasis or peritoneal carcinomatosis. 8. Intestinal obstruction. 9. Existence of microsatellite instability 10. Refusal to participate or to give written consent 11. Impossibility, at the investigator's discretion, to understand the purpose of the study or to comply with its procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2023-05-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (SLE) at 2 years | From the inclusion of the patient in the study to 5 years of follow-up or his death, whichever comes first.
  To determine whether the proposed treatment with neoadjuvant chemotherapy, surgery and complementary chemotherapy increases the disease-free survival (SLE) at 2 years postoperatively, compared with standard treatment, surgery and complementary chemotherapy.

SECONDARY OUTCOMES:
To assess whether neoadjuvant chemotherapy, surgery and complementary chemotherapy increases SLE 5 years postoperatively, compared to standard treatment of surgery and complementary chemotherapy | From the inclusion of the patient in the study to 5 years of follow-up or his death, whichever comes first.
  From the inclusion of the patient in the study to 5 years of follow-up or his death, whichever comes first.
To evaluate whether neoadjuvant chemotherapy, surgery and complementary chemotherapy increase OS at 2 and 5 years postoperatively, in comparison with standard treatment of surgery and complementary chemotherapy. | From the inclusion of the patient in the study to 5 years of follow-up or his death, whichever comes first.
  From the inclusion of the patient in the study to 5 years of follow-up or his death, whichever comes first.
To compare the postoperative morbidity and mortality of the neoadjuvant treatment in relation to the standard treatment | From the inclusion of the patient in the study to 5 years of follow-up or his death, whichever comes first.
  From the inclusion of the patient in the study to 5 years of follow-up or his death, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: JORGE ARREDONDO, DR., Principal Investigator — COMPLEJO ASISTENCIAL UNIVERSITARIO DE LEON
Locations (1):
- Complejo Asistencial Universitario de Leon, León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arredondo J, Almeida A, Castanon C, Sanchez C, Villafane A, Tejedor P, Simo V, Baixauli J, Rodriguez J, Pastor C. The ELECLA trial: A multicentre randomised control trial on outcomes of neoadjuvant treatment on locally advanced colon cancer. Colorectal Dis. 2024 Apr;26(4):745-753. doi: 10.1111/codi.16908. Epub 2024 Feb 16. PMID 38362850
- See also: Spanish Registry of Clinical Studies — http://reec.aemps.es/reec/public/web.html